CLINICAL TRIAL: NCT05621681
Title: Postoperative Pain Assessment Following Unintentional Bioceramic Sealer Extrusion
Brief Title: This Prospective Study Has 2 Objectives: First, to Assess the Post-obturation Pain Utilizing Bioceramic Sealer and One Cone Technique. Second, to Compare the Intensity of Post-obturation Pain Following Unintentional Sealer Extrusion
Status: Completed | Type: Observational
Sponsor: Abdulaziz Abdulmunim Alabdulmunim (Other)
Responsible Party: Sponsor-Investigator, Abdulaziz Abdulmunim Alabdulmunim, Intern, Qassim University
Organization: Qassim University (Other)
Other Study IDs: Abdulaziz Abdulmunim
Record Dates: First submitted 2022-11-05; First posted 2022-11-18 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-04

CONDITIONS: Pain, Postoperative; Endodontic Overfill
Keywords: Sealer extrusion; Postoperative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Root canal treatment is essential step to eliminate pain and preserve tooth structures. However, errors could happen unintentionally such as ledge, perforation and sealer extrusion.

Pain through an endodontic treatment is one of the elements that most of the patients seek treatment to be relived.

One the current systemic review analyzed the pain after root canal treatment could be up to half the patients.

The purpose of this study is to evaluate and record the postoperative pain among patients who are undergoing root canal treatment.

ELIGIBILITY:
"Inclusion Criteria":

* Primary root canal
* Asymptomatic tooth with or without apical radiolucency
* Patient older than 18 and younger than 70
* American Society of Anesthesiology (ASA) Class I or II

"Exclusion Criteria":

* Patient with preoperative pain
* Periodontal probing more than 5mm
* When patency could not be achieved
* pregnant patient.,
* patients who could not properly follow the instructions for filling the visual analog card (VAS) were excluded.
* Previously treated or initiated

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary dental care
Sampling Method: Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Each patient was given visual assessment scale to analyze the postoperative pain and assessing the change in different time intervals (6 hours,24 hours,2 days,3days and 4 days) | Five times intervals were recorded at the following: 6 hours following the treatment,1 day,2days,3days and 4 days
  Visual analogue card scales contains numbers range from 0-10 1-3 indicates mild pain, while 4-6 suggests moderate pain and 7-10 specify sever pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Abdulaziz Abdulmunim, Buraidah, Al-Qassim Region, Saudi Arabia